CLINICAL TRIAL: NCT03014245
Title: Circulating Melatonin and 6-hydroxymelatonin Levels During Pregnancy
Brief Title: Melatonin in Pregnancy Compared to Non-pregnant
Acronym: MEL-P
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2/08/16
Record Dates: First submitted 2016-12-12; First posted 2017-01-09 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-01

CONDITIONS: Pregnancy Transient Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant: Normal pregnant women (first baby) singleton
- Control: Non pregnant healthy women

SUMMARY:
Melatonin is well known for its role in the sleep-wake cycle but it is less well known as an effective antioxidant. It has been reported to be synthesised in the placenta and may have both receptor mediated and non-receptor mediated protective functions during pregnancy. Severe pre-eclampsia has been reported to be associated with low levels of melatonin in the placenta although it is not known if the placental melatonin contributes to circulating levels. There is little reported on the circulating levels of melatonin or oxidative stress at different stages of normal pregnancy. More information on the role of melatonin and metabolism of melatonin in pregnancy as well as any significant association with adverse pregnancy outcomes would inform planning of larger research studies to investigate the potential role for melatonin as a biomarker for obstetric disease and potentially as a therapeutic agent in future.

This observational pilot study aims to measure serum melatonin levels and 6-hydroxymelatonin sulphate (the major metabolite of melatonin) during each trimester of pregnancy.

DETAILED DESCRIPTION:
Melatonin, a substance produced by the pineal gland, is well known for its role in the sleep-wake cycle but it is less well known as an effective antioxidant. It is able to access all parts of the cell, and can cross the blood-brain and placental barrier. Melatonin has been reported to be synthesised in the placenta and may have both receptor mediated and non-receptor mediated protective functions during pregnancy. Severe pre-eclampsia has been reported to be associated with low levels of melatonin in the placenta although it is not known if the placental melatonin contributes to circulating levels. Despite this, melatonin levels have been proposed as a biomarker of pre-eclampsia. A further study suggested pregnant women with hypertensive or diabetic conditions had lower melatonin levels and less circadian variation, again suggesting the potential protective role melatonin may have during pregnancy. Due to its antioxidant effects melatonin has also been proposed as a protective substance for women undergoing assisted reproduction techniques.

Rationale for study There is little reported on the circulating levels of melatonin or oxidative stress at different stages of normal pregnancy. More information on the role of melatonin and metabolism of melatonin in pregnancy as well as any significant association with adverse pregnancy outcomes would inform planning of larger research studies to investigate the potential role for melatonin as a bio-marker for obstetric disease and potentially as a therapeutic agent in future.

This observational pilot study aims to measure serum melatonin levels and 6-hydroxymelatonin sulphate (the major metabolite of melatonin) during each trimester of pregnancy.

STUDY OBJECTIVES Objectives Primary Objective To determine if serum melatonin and 6-hydroxymelatonin sulphate levels differ in each trimester of pregnancy and how these compare to non-pregnant women Secondary Objectives

1. To determine level of oxidative stress at time of serum sample by measuring lipid peroxide levels
2. To explore whether levels of serum melatonin and 6-hydroxymelatonin sulphate vary in women who develop antenatal complications (pre-eclampsia or hypertensive diseases of pregnancy, preterm labour or gestational diabetes)

OUTCOMES Primary Outcome Serum melatonin and 6-hydroxymelatonin sulphate levels Secondary Outcomes

1. Level of oxidative stress at time of sampling (lipid peroxide levels)
2. Outcome of pregnancy (live birth or not, development of preeclampsia / hypertensive disease of pregnancy, gestational diabetes or preterm labor.

STUDY DESIGN Study Description

Twenty healthy women in their first pregnancy will be recruited at their first antenatal (scan) visit at 11-13 weeks gestation. Recruitment will continue throughout the medical student's allocated project time period to allow recruitment of as many women as possible, but at least twenty pregnant women. A venous blood sample to measure serum melatonin and 6-hydroxymelatonin sulphate levels will be obtained using aseptic technique. Sampling, when possible, will be carried out at the same time as for routine clinical screening. The first blood sample will be done at 11-13 weeks gestation (first trimester) and could be done along with routine antenatal screening blood tests. A second blood sample will be taken when women attend for their detailed ultrasound scan at approximately 20 weeks (2nd trimester). The participant may not need other routine blood tests at this time, therefore this blood sample would only be for the purpose of the study.

A third and final blood sample will be obtained at around 28 weeks gestation (third trimester). This could be done at the routine 28 week appointment with the participant's community midwife when routine pregnancy blood tests will already be undertaken. Consent will be sought from the participant to contact the applicable community midwife to arrange to attend the midwifery appointment at around 28 weeks. The third blood sample will be taken either at Aberdeen Maternity Hospital or at the participant's GP practice depending on preference and convenience of appointment location for the participant and community midwife. The researchers will not contact the participant directly. If the woman is attending the obstetric antenatal clinic at that gestation the blood sample could alternatively be obtained there along with the routine antenatal screening blood tests.

Non-pregnant controls will be recruited by advertising using posters around the University of Aberdeen/Aberdeen Royal Infirmary campus, aiming for 20 non pregnant women, aged between 16 and 45 to have blood samples taken for serum melatonin and 6-hydroxy-melatonin sulphate levels. Samples will be taken at the same time of day and year as pregnant subjects to account for any seasonal effects.

Serum melatonin will be measured using liquid chromatography-tandem mass spectrometry and 6-hydroxymelatonin sulphate will be measured using enzyme immunoassay. Lipid peroxides will be measured using a colorimetric assay.

Written informed consent will be obtained from all participants. Women will be asked for their age, body mass index, gestation stage, smoking status, name of their community midwife and a series of screening questions to determine eligibility according to inclusion criteria. Once recruited, an anonymous code will be assigned and all data will be kept separately from identifiable information.

ELIGIBILITY:
Inclusion Criteria:

Pregnant subjects

* Primigravid women (in their first pregnancy)
* Singleton pregnancy
* Aged 16-45
* Taking no regular medication other than pregnancy related vitamins or supplements
* First trimester (FVS) ultrasound scan reported as normal

Non pregnant subjects

* Non pregnant women
* Aged 16-45
* No chronic health issues and not taking any medication

Exclusion Criteria:

Pregnant subjects

* Pregnancy non-viable on scan
* Twins or higher multiple pregnancies
* Outside age range
* Diabetes or pre-existing hypertension, chronic kidney disease or known autoimmune disorder

Non pregnant subjects

* Male
* Outside age range
* Chronic health complaint/taking medication
* Recent blood donation over 1 unit

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy women pregnant with first baby (singleton) presenting for first trimester scan and healthy non-pregnant women of child bearing age.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Change in melatonin and 6-hydroxymelatonin levels during pregnancy | Values up to 40 weeks
  Do serum melatonin and 6-hydroxymelatonin sulphate levels differ in each trimester of pregnancy? Levels during each trimester will be compared.

SECONDARY OUTCOMES:
Change in lipid peroxide levels during pregnancy | Values up to 40 weeks
  Does oxidative stress (lipid peroxide levels) vary in each trimester. Levels during each trimester will be compared.
Relationship between melatonin and 6-hydroxymelatonin levels and duration of pregnancy. | Up to 40 weeks
  What is melatonin status in women who deliver at different gestation (in weeks).
Relationship between melatonin and 6-hydroxymelatonin levels with different types of delivery. | Up to 40 weeks
  What is melatonin status in women with different labours (induced, spontaneous or planned caesarean section)
Relationship between melatonin and 6-hydroxymelatonin levels and pre-eclampsia | Up to 40 weeks
  What is melatonin status in women who had pre-eclampsia ( as yes/no) and those who did not.
Relationship between melatonin and 6-hydroxymelatonin levels and gestational diabetes | Up to 40 weeks
  What is melatonin status in women who had gestational diabetes ( as yes/no) compared to those who did not.
Melatonin and 6-hydroxymelatonin levels in pregnancy compared to non pregnant | Up to 40 weeks
  Is melatonin status at any time during pregnancy different to that in healthy non pregnant women? :Levels of melatonin and 6-hydroxymelatonin in non-pregnant women will be compared with levels in pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Maternity Hospital (NHS Grampian), Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No